CLINICAL TRIAL: NCT01116921
Title: Laryngeal Mask Airway (LMA) for Surfactant Administration in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1004M81177
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Respiratory Distress Syndrome
Keywords: laryngeal mask airway; surfactant; respiratory distress syndrome; neonate
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure; Laryngeal Masks; Pulmonary Surfactants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nCPAP Control Group (Active Comparator): Infants in the Control Group were maintained continuously on nasal CPAP 6 cm H2O with no surfactant administered.
  Interventions: Device: Nasal continuous positive airway pressure (nCPAP)
- LMA Group (Experimental): Once proper placement of the LMA was achieved, surfactant (Curosurf®, 2.5 ml/kg, Chiesi USA, Inc., Cary, NC) was administered. The LMA cuff was then deflated, LMA removed and the infant placed back on nasal CPAP 6 cm H2O.
  Interventions: Device: Nasal continuous positive airway pressure (nCPAP); Device: Laryngeal Mask Airway (LMA) to deliver surfactant; Drug: Surfactants, Pulmonary

INTERVENTIONS:
Device: Nasal continuous positive airway pressure (nCPAP) — nCPAP equipment used in the trial will be the standard hospital equipment used in the NICU.
Device: Laryngeal Mask Airway (LMA) to deliver surfactant — Laryngeal Mask Airway (LMA Unique-Size 1, The Laryngeal Mask Company Limited, San Diego, CA)
  Arms: LMA Group
Drug: Surfactants, Pulmonary — Curosurf®, Chiesi USA, Inc., Cary, NC
  Arms: LMA Group

SUMMARY:
The primary objective of this research is to compare the need for intubation and mechanical ventilation in the first seven days of life for infants with respiratory distress syndrome (RDS) on nasal continuous positive airway pressure (nCPAP) who receive surfactant via a Laryngeal Mask Airway (LMA) with those who are maintained on nCPAP and do not receive surfactant.

DETAILED DESCRIPTION:
Secondary outcomes were total number of hours on mechanical ventilation, CPAP and supplemental oxygen during the first 7 days of life and for the entire hospitalization. Other secondary outcomes were number of surfactant doses, incidence of pulmonary air leak, survival until discharge, chronic lung disease (defined as need for oxygen at 36 weeks PMA), oxygen requirement at discharge, severe intraventricular hemorrhage (Grade 3/4), and periventricular leukomalacia.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at time of enrollment 28 0/7 to 35 6/7 weeks postmenstrual age
* Age less than or equal to 36 hours old
* On nCPAP 6 with supplemental oxygen requirement (Fi02 greater than or equal to 30%) for greater than or equal to 30 minutes (to maintain Sa02 between 88-92%)
* Chest radiograph and clinical presentation consistent with respiratory distress syndrome (tachypnea, retractions, nasal flaring, and/or grunting

Exclusion Criteria:

* Prior mechanical ventilation or surfactant administration
* Major congenital anomaly
* Abnormality of the airway
* Respiratory distress secondary to an etiology other than respiratory distress syndrome (pneumothorax, meconium aspiration syndrome, pneumonia, hypoxic-ischemic encephalopathy)
* Apgar score < 5 at 5 minutes of age

Max Age: 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari D Roberts, M.D., Study Chair — University of Minnesota Masonic Children's Hospital; Sijani Tipnis, M.D., Principal Investigator — University of California, San Diego; Andrea L Lampland, M.D., Principal Investigator — St Paul Children's Hospital; Allen Merritt, M.D., Principal Investigator — Loma Linda University; Erin Stepka, M.D., Principal Investigator — Maple Grove Hospital and North Memorial Hospital; Julie Kessel, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (7):
- United States (7):
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California- San Diego Medical Center, San Diego, California
  - Maple Grove Hospital, Maple Grove, Minnesota
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - North Memorial Hospital, Robbinsdale, Minnesota
  - St Paul Children's Hospital, Saint Paul, Minnesota
  - University of Wisconsin- Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wanous AA, Brown R, Rudser KD, Roberts KD. Comparison of laryngeal mask airway and endotracheal tube placement in neonates. J Perinatol. 2024 Feb;44(2):239-243. doi: 10.1038/s41372-023-01818-x. Epub 2023 Nov 2. PMID 37919512
- [Derived] Roberts K, Wanous A, Brown R, Rudser K. Comparison of Laryngeal Mask Airway and Endotracheal Tube Placement in Neonates. Res Sq [Preprint]. 2023 Jul 13:rs.3.rs-3136331. doi: 10.21203/rs.3.rs-3136331/v1. PMID 37503152
- [Derived] Roberts KD, Brown R, Lampland AL, Leone TA, Rudser KD, Finer NN, Rich WD, Merritt TA, Czynski AJ, Kessel JM, Tipnis SM, Stepka EC, Mammel MC. Laryngeal Mask Airway for Surfactant Administration in Neonates: A Randomized, Controlled Trial. J Pediatr. 2018 Feb;193:40-46.e1. doi: 10.1016/j.jpeds.2017.09.068. Epub 2017 Nov 22. PMID 29174079

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | nCPAP Control Group | LMA Group
Started | 53 | 50
Completed | 53 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nCPAP Control Group | LMA Group | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 50 | 103
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age
  weeks | 32.86 (1.86) | 32.71 (1.86) | 32.71 (1.86)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 35 | 30 | 65
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Need for Intubation and Mechanical Ventilation in the First Seven Days of Life.
Description: "Treatment Failure" criteria were the same for both groups. "Treatment Failure" required two of the following: 1) FiO2 >40% for longer than 30 minutes (to maintain SaO2 88-92%), 2) PCO2 >65mmHg on ABG/CBG or >70 on VBG, or 3) pH<7.22 on ABG/CBG/VBG or one of the following: 1) recurrent or severe apnea, 2) hemodynamic instability requiring pressors, 3) repeat surfactant dose at appropriate time with FiO2 >40%, or 4) deemed necessary by medical provider.
Time Frame: Seven days
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
Participants | 34 | 19
Statistical Analysis 1: Comparison: nCPAP Control Group vs LMA Group; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.13 to 0.70]

2. Secondary Outcome: Duration of CPAP Therapy
Time Frame: During first seven days of life
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
hours | 50 (41) | 56 (35)

3. Secondary Outcome: Duration of Oxygen Therapy
Time Frame: During first seven days of life
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
hours | 55 (41) | 56 (45)

4. Secondary Outcome: Incidence of Pulmonary Airleaks
Time Frame: First 7 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
Participants | 5 | 4

5. Secondary Outcome: Incidence of Severe IVH or PVL
Time Frame: During hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
Participants | 0 | 0

6. Secondary Outcome: Incidence of Chronic Lung Disease
Time Frame: Measured at hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | nCPAP Control Group | LMA Group
Number analyzed (Participants) | 53 | 50
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | nCPAP Control Group | LMA Group
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 5/53 | 4/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nCPAP Control Group (N=53) | LMA Group (N=50)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No